CLINICAL TRIAL: NCT03738319
Title: Non-coding RNA in the Exosome of the Epithelia Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EOC-EXOSOME
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: High Grade Serous Carcinoma; Ovarian Cancer; Exosomes; Prognosis; Early Diagnosis
MeSH Terms: conditions — Ovarian Neoplasms; Disease | interventions — RNA, Long Noncoding

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — An 8 ml peripheral venous blood will be collected from the participants before and after interventions (i.e. surgery and/or chemotherapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HGSOC group: This group includes patients of high grade serous ovarian cancer (HGSOC).
  Interventions: Genetic: Sequencing of miRNA/lncRNA
- Control group: This group includes patients of benign gynecologic diseases as control.
  Interventions: Genetic: Sequencing of miRNA/lncRNA

INTERVENTIONS:
Genetic: Sequencing of miRNA/lncRNA — Next generation sequencing of micro-RNA (miRNA) and long non-coding RNA (lncRNA)

SUMMARY:
This study aims to analyze the expression of micro-RNA (miRNA) and long non-coding RNA (lncRNA) by next-generation sequencing in patients with high grade serous ovarian cancer (HGSOC) and benign gynecologic diseases. The candidate miRNA/lncRNA will be validated as biomarker for the detection and prognosis of HGSOC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary high grade serous ovarian cancer
* Willing to accepted debulking surgeries and adjuvant chemotherapy
* Good performance status
* Aged 18 years or older
* Signed an approved informed consents

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be 20 patients of high grade serous ovarian cancer (HGSOC) and 20 patients with benign gynecologic diseases, whose data will be applied for construction of diagnostic model of miRNA/lncRNA from exosome. There will be 120 patients suspected of HGSOC, whose data will be applied for validation of such diagnosis model.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-11-23 (Estimated); Study Completion 2019-11-23 (Estimated)

PRIMARY OUTCOMES:
Differential expression of miRNA/lncRNA | One year
  Differential expression of micro-RNA (miRNA) and long non-coding RNA (lncRNA) will be compared between HGSOC group and control group, hence candidate miRNA/lncRNA will be validated as biomarker for the detection and prognosis of HGSOC.

SECONDARY OUTCOMES:
Progression-free survival | Five years
  The progression-free survival of HGSOC patients will be compared between differential expressed candidate miRNA/lncRNA after they have completed debulking surgeries and adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All data will be available to all researchers.
Supporting Information: CSR
Time Frame: All data will be available to all researchers once related papers have been accepted publicly, and will be available for ever.